CLINICAL TRIAL: NCT01977144
Title: Screening of Low Responders for Aneuploidy to Improve Reproductive Efficiency
Acronym: Solaire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RMA1-13-290; RMA-2013-03 (Other: RMANJ)
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Infertility
Keywords: Single Embryo Transfer; Double Embryo Transfer; CCS (Comprehensive Chromosome Screening); Aneuploidy; Low Responders
MeSH Terms: conditions — Infertility; Aneuploidy | interventions — Prostaglandins D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Embryo Transfer with CCS (Other): Patients will have either a single or double embryo transfer with CCS tested embryos
  Interventions: Other: Comprehensive Chromosomal Screening
- Embryo Transfer without CCS (No Intervention): Patients in this group will not have CCS performed on their embryo(s)

INTERVENTIONS:
Other: Comprehensive Chromosomal Screening
  Other Names: PGD
  Arms: Embryo Transfer with CCS

SUMMARY:
The purpose of this study is to assess the impact of Comprehensive Chromosome Screening(CCS) on patients with low ovarian reserve in an effort to improve success during in vitro fertilization and decrease the time to successful pregnancy.

DETAILED DESCRIPTION:
Patients will undergo a stimulated IVF cycle culminating with an ultrasound guided egg retrieval procedure and either a fresh or frozen embryo transfer as clinically appropriate and without regard to study. All embryology laboratory procedures will be conducted per routine. Once the embryo(s) have reached the blastocyst stage of development patients will be randomized into either the study group or the control group. The SOLAIRE Trial is "blinded" which means neither patients nor the RMANJ study doctor/staff will know to which group the embryos were randomized. The study group will have their embryo(s) biopsied for CCS on day 5, if appropriate, for a fresh day 6 embryo transfer. The control group will not have CCS testing performed on their embryo(s) and may proceed with a fresh or frozen embryo transfer as clinically appropriate. The maximum amount of embryos that can be transferred is two per RMANJ protocol. All post-transfer care and pregnancy monitoring will be identical and per routine protocol regardless of study participation.

ELIGIBILITY:
Inclusion Criteria:

* Age of female partner < 43 y/o AMH < 1.1 OR BAFC < 8 (within previous year) Male must have >100,000 motile sperm BMI < 32

Exclusion Criteria:

* Diagnosis of endometrial insufficiency Use of oocyte donor/gestational carriers Use of surgical sperm or DNA Banking Communicating hydosalpinges (HSG) Single gene disorders or sex selection Participation in another study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Delivery rate | 2 years

SECONDARY OUTCOMES:
pregnancy rate per ET | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, HCLD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

REFERENCES:
- [Derived] Cornelisse S, Zagers M, Kostova E, Fleischer K, van Wely M, Mastenbroek S. Preimplantation genetic testing for aneuploidies (abnormal number of chromosomes) in in vitro fertilisation. Cochrane Database Syst Rev. 2020 Sep 8;9(9):CD005291. doi: 10.1002/14651858.CD005291.pub3. PMID 32898291